CLINICAL TRIAL: NCT06366750
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Barzolvolimab (CDX-0159) in Patients With Prurigo Nodularis
Brief Title: A Study of Barzolvolimab in Patients With Prurigo Nodularis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDX0159-10; 2023-510279-80-00 (Other: EU CT)
Record Dates: First submitted 2024-03-27; First posted 2024-04-16 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Prurigo Nodularis
Keywords: barzolvolimab; PN; CDX-0159

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Barzolvolimab 450 mg, then 150 mg Q4W (Experimental): 450 mg subcutaneous administration loading dose on Day 1 followed by 150 mg subcutaneous administration every 4 weeks, starting on Week 4, to Week 24.
  Interventions: Biological: barzolvolimab
- Barzolvolimab 450 mg, then 300 mg Q4W (Experimental): 450 mg subcutaneous administration loading dose on Day 1 followed by 300 mg subcutaneous administration every 4 weeks, starting on Week 4, to Week 24.
  Interventions: Biological: barzolvolimab
- Placebo (Placebo Comparator): Matching placebo subcutaneous administration every 4 weeks, starting on Week 4, to Week 24.
  Interventions: Other: Matching Placebo

INTERVENTIONS:
Biological: barzolvolimab — subcutaneous administration
  Arms: Barzolvolimab 450 mg, then 150 mg Q4W; Barzolvolimab 450 mg, then 300 mg Q4W
Other: Matching Placebo — subcutaneous administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of barzolvolimab in adults with prurigo nodularis.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy and safety of barzolvolimab (CDX-0159) in adults with prurigo nodularis.

There is a screening period of approximately 28 days, a 24-week double-blind treatment period and a 16-week follow-up period after treatment. Participants will be randomly assigned on a 1:1:1 ratio to receive barzolvolimab (CDX-0159) by subcutaneous injections of 150 mg every 4 weeks (Q4W) after an initial loading dose of 450 mg, 300 mg Q4W after an initial loading dose of 450 mg, or placebo Q4W.

Following the completion of the treatment period, participants may enter an open label extension portion of the study if they are eligible.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males and females, ≥18 years of age.
2. Diagnosis of Prurigo Nodularis by a dermatologist at least 3 months prior to Screening with:

   1. At least 20 PN nodules with bilateral distribution on both arms and/or both legs and/or both sides of the trunk at screening.
   2. An Investigators Global Assessment for stage of chronic nodular prurigo (IGA-CNPG-S) score for PN ≥ 3 at screening and Baseline (Day 1).
3. Severe itch, defined as the mean of the daily worst itch NRS (WI-NRS) score of ≥ 7 during the 7-day period immediately prior to initiation of study treatment.
4. Documented history of inadequate response to prescription topical medications or for whom topical medications are medically inadvisable.
5. Willing to apply a topical moisturizer (emollient) once or twice a day throughout the study.
6. Both males and females of child-bearing potential must agree to use highly effective contraceptives during the study and for 150 days afterwards after treatment.
7. Willing and able to complete a daily symptom electronic diary for the duration of the study and adhere to the study visit schedule.

Key Exclusion Criteria

1. PN due to neuropathy, psychiatric disorders or medications.
2. Unilateral PN lesions limited to small area on one side of the body (e.g., only one arm affected).
3. Active unstable pruritic skin conditions in addition to PN.
4. Documented atopic dermatitis (moderate to severe) within 6 months before the start of screening.
5. Females who are pregnant or nursing.
6. Known hepatitis B or hepatitis C infection or active COVID-19 infection.
7. Vaccination with a live vaccine within 2 months prior to study drug administration (subjects must agree to avoid vaccination during the study and for four months thereafter). NOTE: Inactivated vaccines are allowed such as seasonal influenza for injection. COVID-19 vaccination is allowed.
8. History of anaphylaxis.
9. Prior receipt of barzolvolimab

There are additional criteria that your study doctor will review with you to confirm you are eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2024-04-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with improvement in Worst Itch Numeric Rating Scale (WI-NRS) by ≥ 4 from baseline to Week 12. | From Day 1 (first dose) to Day 85 (week 12)
  WI-NRS is a validated measure of itch severity. Participants are asked daily to rate the intensity of their worst pruritis (itch) over the past 24 hours using an 11-point scale ranging from 0= no itch to 10= worst imaginable itch. Higher scores indicate more severity.

SECONDARY OUTCOMES:
Proportion of participants with improvement in WI-NRS by ≥ 4 from baseline to Week 4. | From Day 1 (first dose) to Week 4
  WI-NRS is a validated measure of itch severity. Participants are asked daily to rate the intensity of their worst pruritis (itch) over the past 24 hours using an 11-point scale ranging from 0= no itch to 10= worst imaginable itch. Higher scores indicate more severity.
Proportion of participants with improvement in WI-NRS by ≥ 4 from baseline to Week 24. | From Day 1 (first dose) to Week 24
  WI-NRS is a validated measure of itch severity. Participants are asked daily to rate the intensity of their worst pruritis (itch) over the past 24 hours using an 11-point scale ranging from 0= no itch to 10= worst imaginable itch. Higher scores indicate more severity.
Proportion of participants with improvement in WI-NRS by ≥ 4 from baseline to Day 169 (week 24). | From Day 1 (first dose) to Day 169 (week 24)
  WI-NRS is a validated measure of itch severity. Participants are asked daily to rate the intensity of their worst pruritis (itch) over the past 24 hours using an 11-point scale ranging from 0= no itch to 10= worst imaginable itch. Higher scores indicate more severity.
Proportion of participants with Investigator Global Assessment for stage of chronic nodular prurigo score (IGA-CNPG-S) of 0 or 1 at Weeks 4, 12 and 24. | From Day 1 (first dose) to Day 169 (week 24)
  The IGA-CNPG-S is an instrument used to assess the overall number of PN lesions at a given timepoint, as determined by the investigator. It consists of a 5-point scale ranging from 0 to 4 where 0= clear, 1= almost clear, 2= mild, 3= moderate, and 4= severe. Higher scores indicate severe PN. In this outcome measure, percentage of participants with an IGA-CNPG-S score of either 0 or 1 at Weeks 4, 12 and 24 will be reported.
Proportion of participants with improvement in both WI-NRS by ≥ 4 from baseline and IGA-CNPG-S score of 0 or 1 at Weeks 4, 12 and 24. | From Day 1 (first dose) to Day 169 (week 24)
  WI-NRS is a validated measure of itch severity. Participants are asked daily to rate the intensity of their worst pruritis (itch) over the past 24 hours using an 11-point scale ranging from 0 = no itch to 10 =worst imaginable itch. Higher scores indicate more severity.
  The Investigator Global Assessment for stage of chronic nodular prurigo (IGA-CNPG-S) is an instrument used to assess the overall number of PN lesions at a given timepoint, as determined by the investigator. It consists of a 5-point scale ranging from 0 to 4 where 0= clear, 1= almost clear, 2= mild, 3= moderate, and 4= severe. Higher scores indicate severe PN.
  Percentage of participants who achieve both an improvement in WI-NRS and an improvement in IGA-CNPG-S will be reported in this outcome.
Proportion of participants with Investigator Global Assessment for activity of chronic prurigo (IGA-CPG-A) score of 0 or 1 at Weeks 4, 12 and 24. | From Day 1 (first dose) to Day 169 (week 24)
  The IGA-CPG-A is an instrument used to assess the overall activity of PN lesions at a given time point, as determined by the investigator. It consists of a 5-point scale ranging from 0-4 where 0= clear (0% lesions showing excoriations/crusts), 1= almost clear (1-10% lesions showing excoriations/crusts), 2= Mild (11-25% lesions showing excoriations/crusts), 3= moderate (26-75% lesions showing excoriations/crusts), 4= severe (76-100% lesions showing excoriations/crusts). Higher scores indicate severe PN. In this outcome measure, percentage of participants with an IGA-CPG-A score of either 0 (clear) or 1 (almost clear) at Weeks 4,12 and 24 will be reported.
Absolute change from baseline in WI-NRS at Weeks 4, 12 and 24. | From Day 1 (first dose) to Day 169 (week 24)
  WI-NRS is a validated measure of itch severity. Participants are asked daily to rate the intensity of their worst pruritis (itch) over the past 24 hours using an 11-point scale ranging from 0= no itch to 10= worst imaginable itch. Higher scores indicate more severity.
Percentage change from baseline in WI-NRS at Weeks 4, 12 and 24. | From Day 1 (first dose) to Day 169 (week 24)
  WI-NRS is a validated measure of itch severity. Participants are asked daily to rate the intensity of their worst pruritis (itch) over the past 24 hours using an 11-point scale ranging from 0= no itch to 10= worst imaginable itch. Higher scores indicate more severity.
Absolute change from baseline in Sleep Quality Numerical Rating Scale (SQ-NRS) at Weeks 4, 12 and 24. | From Day 1 (first dose) to Day 169 (week 24)
  SQ-NRS is an assessment where participants rate their sleep during the past 24 hours as a score ranging from 0= best possible sleep to 10= worst possible sleep. Higher scores indicate more severity.
Percentage change from baseline in SQ-NRS at Weeks 4, 12 and 24. | From Day 1 (first dose) to Day 169 (week 24)
  SQ-NRS is an assessment where participants rate their sleep during the past 24 hours as a score ranging from 0= best possible sleep to 10= worst possible sleep. Higher scores indicate more severity.
Absolute change from baseline in Worst Pain Numerical Rating Scale (WP-NRS) at Weeks 4, 12 and 24. | From Day 1 (first dose) to Day 169 (week 24)
  WP-NRS is used to measure skin pain intensity. Participants are asked to rate their worst pain during the past 24 hours as a score ranging from 0= no pain to 10= worst imaginable pain. Higher scores indicate more severity.
Percentage change from baseline in WP-NRS at Weeks 4, 12 and 24. | From Day 1 (first dose) to Day 169 (week 24)
  Worst Pain Numerical Rating Scale (WP-NRS) is used to measure skin pain intensity. Participants are asked to rate their worst pain during the past 24 hours as a score ranging from 0= no pain to 10= worst imaginable pain. Higher scores indicate more severity.
Absolute change from baseline in Patient-Reported Outcomes Measurement Information System Fatigue - Short Form 7b Daily (PROMIS Fatigue-SF Daily) at Weeks 4, 12 and 24. | From Day 1 (first dose) to Day 169 (week 24)
  PROMIS Fatigue-SF Daily is an assessment where participants rate their fatigue on a daily basis by responding to 7 questions. Each question is based on a 5-point scale ranging from 1= never to 5= always.
Percentage change from baseline in PROMIS Fatigue-SF Daily at Weeks 4, 12 and 24. | From Day 1 (first dose) to Day 169 (week 24)
  Patient-Reported Outcomes Measurement Information System Fatigue - Short Form 7b Daily (PROMIS Fatigue-SF Daily) is an assessment where participants rate their fatigue on a daily basis by responding to 7 questions. Each question is based on a 5-point scale ranging from 1= never to 5= always.
Absolute change from baseline in Dermatology Life Quality Index (DLQI) at Weeks 4, 12 and 24. | From Day 1 (first dose) to Day 169 (week 24)
  The DLQI is a self-administered, dermatology-specific quality of life (QoL) questionnaire that consists of 10 questions concerning participants' perception of the impact of their skin disease on different aspects of their QoL (symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment) over the previous week. The DLQI score ranges from 0= no effect on the participant's life to 30= extremely large effect on the participant's life.
Percentage change from baseline in Dermatology Life Quality Index (DLQI) at Weeks 4, 12 and 24. | From Day 1 (first dose) to Day 169 (week 24)
  The DLQI is a self-administered, dermatology-specific quality of life (QoL) questionnaire that consists of 10 questions concerning participants' perception of the impact of their skin disease on different aspects of their QoL (symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment) over the previous week. The DLQI score ranges from 0= no effect on the participant's life to 30= extremely large effect on the participant's life.
Proportion of participants with WI-NRS score < 2 at Weeks 4, 12 and 24. | From Day 1 (first dose) to Day 169 (week 24)
  WI-NRS is a validated measure of itch severity. Participants are asked daily to rate the intensity of their worst pruritis (itch) over the past 24 hours using an 11-point scale ranging from 0 = no itch to 10 = worst imaginable itch. Higher scores indicate more severity. In this outcome measure, the proportion of participants with an improvement (reduction) in WI-NRS to a score of < 2 at Weeks 4, 12 and 24, will be reported.
Proportion of participants with improvement in SQ-NRS by ≥ 4 from baseline to Week 4, 12 and 24. | From Day 1 (first dose) to Day 169 (week 24)
  Sleep Quality Numerical Rating Scale (SQ-NRS) is an assessment where participants rate their sleep during the past 24 hours as a score ranging from 0 = best possible sleep to 10 = worst possible sleep. Higher scores indicate more severity.
Proportion of participants with improvement in WP-NRS by ≥ 4 from baseline to Weeks 4, 12 and 24. | From Day 1 (first dose) to Day 169 (week 24)
  Worst Pain Numerical Rating Scale (WP-NRS) is used to measure skin pain intensity. Participants are asked to rate their worst pain during the past 24 hours as a score ranging from 0 = no pain to 10 = worst imaginable pain. Higher scores indicate more severity.
Proportion of participants with improvement of ≥ 4 in DLQI from baseline to Weeks 4, 12 and 24. | From Day 1 (first dose) to Day 169 (week 24)
  The DLQI is a self-administered, dermatology-specific quality of life (QoL) questionnaire that consists of 10 questions concerning participants' perception of the impact of their skin disease on different aspects of their QoL (symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment) over the previous week. The DLQI score ranges from 0= no effect on the participant's life to 30= extremely large effect on the participant's life. Proportion of participants with improvement in DLQI scores of ≥ 4 points from baseline to Weeks 4,12 and 24 will be reported.
Proportion of participants achieving DLQI score of 0 or 1 at Weeks 4, 12 and 24. | From Day 1 (first dose) to Day 169 (week 24)
  The DLQI is a self-administered, dermatology-specific quality of life (QoL) questionnaire that consists of 10 questions concerning participants' perception of the impact of their skin disease on different aspects of their QoL (symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment) over the previous week. The DLQI score ranges from 0= no effect on the participant's life to 30= extremely large effect on the participant's life. Proportion of participants achieving DLQI scores of 0 or 1 at Weeks 4,12 and 24 will be reported.
Absolute change from baseline in PGIS, PGIS-SD, PGIC and PGIC-SD. | From Day 1 (first dose) to Day 169 (week 24)
  Patient Global Impression of Severity of Disease (PGIS) is an assessment where participants rate the severity in their PN. Patient Global Impression of Severity of Sleep Disturbance (PGIS-SD) is an assessment where participants rate the severity of their sleep disturbance. PGIS and PGIS-SD are gauged on a scale ranging from 0= none to 4= very severe.
  Patient Global Impression of Change of Disease (PGIC) is an assessment where participants rate the change in their PN. Patient Global Impression of Change of Sleep Disturbance (PGIC-SD) is an assessment where the participants rate the change in their sleep disturbance. PGIC and PGIC-SD are gauged on a scale of 1= Much better to 5= Much worse. Participants will be asked to provide this rating in comparison to just before the participant starts taking study treatment.
Percentage change from baseline in PGIS, PGIS-SD, PGIC and PGIC-SD at Weeks 4, 12 and 24. | From Day 1 (first dose) to Day 169 (week 24)
  PGIS is an assessment where participants rate the change in their PN. PGIS-SD is an assessment where participants rate the severity of their sleep disturbance. PGIS and PGIS-SD are gauged on a scale ranging from 0= none to 4= very severe.
  PGIC is an assessment where participants rate the change of their PN. PGIC-SD is an assessment where the participants rate the change in their sleep disturbance. PGIC and PGIC-SD are gauged on a scale of 1= Much better to 5= Much worse. Participants will be asked to provide this rating in comparison to just before the participant starts taking study treatment.
Number of participants with Treatment-Emergent Adverse Events (TEAEs) throughout the study. | From Day 1 (first dose) to Day 281 (last follow-up visit)
  An adverse event (AE) is any untoward medical occurrence in a participant administered study treatment and does not have to have a causal relationship with the treatment. TEAEs are defined as AEs that develop, worsen or become serious during the treatment- emergent (TE) period from the first investigational medicinal product (IMP) administration to the last IMP administration.

CONTACTS AND LOCATIONS:
Locations (72):
- United States (37):
  - Total Dermatology, Birmingham, Alabama
  - Cahaba Dermatology Skin Health Center, Birmingham, Alabama
  - Investigate MD, LLC, Scottsdale, Arizona
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Center for Dermatology Clinical Research, Inc, Fremont, California
  - Profound Research LLC, Oceanside, California
  - Empire Clinical Research, Pomona, California
  - University of California San Francisco, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Dermatology Institute & Skin Care Center, Santa Monica, California
  - Focus Clinical Research, West Hills, California
  - Encore Medical Research Boynton Beach, Boynton Beach, Florida
  - Biobrilliance Medical Research Center, Hialeah, Florida
  - Encore Medical Research, Hollywood, Florida
  - Life Arc Research Centers Corp, Miami, Florida
  - University of Miami, Miami, Florida
  - Advanced Clinical Research Institute, Tampa, Florida
  - Encore Medical Research of Weston, Weston, Florida
  - Emory University, Atlanta, Georgia
  - Centricity Research, Columbus, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - MetroMed Clinical Trials, Chicago, Illinois
  - DS Research of Southern Indiana, LLC, Clarksville, Indiana
  - Equity Medical, Bowling Green, Kentucky
  - DS Research of Kentucky, LLC, Louisville, Kentucky
  - Revival Research Institute, LLC, Troy, Michigan
  - Medisearch, LLC, Saint Joseph, Missouri
  - Skin Specialists PC, Omaha, Nebraska
  - University of New Mexico Department of Dermatology, Albuquerque, New Mexico
  - Equity Medical, New York, New York
  - Apex Clinical Research Center - Canton, Canton, Ohio
  - UC Health Physicians Office Dermatology, Cincinnati, Ohio
  - Paddington Testing, PO, Philadelphia, Pennsylvania
  - Columbia Dermatology and Aesthetics, Columbia, South Carolina
  - International Clinical Research - Tennessee LLC, Murfreesboro, Tennessee
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Center for Clinical Studies, Webster, Texas
- Canada (6):
  - Stratica Dermatology, Edmonton, Alberta
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Kingsway Clinical Research, Etobicoke, Ontario
  - Guelph Dermatology Research, Guelph, Ontario
  - Derm Effects, London, Ontario
  - North York Research Inc, Toronto, Ontario
- Croatia (3):
  - Special Hospital Medico, Rijeka
  - University Hospital Center - Rijeka, Rijeka
  - Solmed Clinic, Zagreb
- Germany (10):
  - Universitätsklinikum Augsburg, Augsburg
  - Fachklinik Bad Bentheim, Klinisches Studienzentrum, Bad Bentheim
  - Institut für Allergieforschung (IFA),Charité - Universitätsmedizin Berlin, Berlin
  - Katholisches Klinikum Bochum, Bochum
  - Universitätsklinikum Erlangen - Hautklinik, Erlangen
  - Universitätsklinikum RWTH Aachen- Dermatology, Frankfurt
  - Universtätsklinikum Frankfurt, Klinik für Dermatologie, Venerologie und, Frankfurt
  - University Hospital Heidelberg, Heidelberg
  - Universitätsklinikum Münster (UKM), Münster
  - Universitätsklinikum Tübingen - Hautklinik, Tübingen
- Poland (11):
  - Centrum Nowoczesnych Terapii "Dobry Lekarz", Krakow, Małopolska
  - FutureMeds Gdynia, Gdynia
  - Centrum Medyczne Pratia Katowice, Katowice
  - Gyncentrum sp. z o.o., Katowice
  - Pratia MCM Krakόw, Krakow
  - LUXDERM Specjalistyczny Gabinet, Lublin
  - Uniwersytecki Szpital Kliniczny im. Fryderyka Chopina w Rzeszowie, Rzeszów
  - Clinical /research group Z.o.o., Warsaw
  - Gyncentrum sp. z o.o., NZOZ Gyncentrum - Oddział Warszawa, Warsaw
  - Klinika Ambroziak Dermatologia, Warsaw
  - DERMACEUM Centrum Badan, Wroclaw
- Spain (5):
  - Complexo Hospitalario Universitario de Santiago de Compostela, A Coruña
  - Hospital General Universitario Dr Balmis, ISABIAL, Alicante
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - FutureMeds - Madrid, Madrid
  - FutureMeds - Sevilla, Seville